CLINICAL TRIAL: NCT03120806
Title: Comparative Study Between Interrupted and Continuous Subcuticular Skin Suturing in Women Undergoing Elective Cesarean Section. A Randomized Controlled Trial
Brief Title: Interrupted Versus Continuous Subcuticular Skin Suturing in Elective Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167
Record Dates: First submitted 2017-04-16; First posted 2017-04-19 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Cesarean Section Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continous subcuticular (Active Comparator): skin closed with continous subcuticular mattress suture using non-absorbable polypropylene
  Interventions: Procedure: continuous subcuticular skin closure
- Interrupted subcuticular (Active Comparator): skin closed with interrupted subcuticular mattress suture using non-absorbable polypropylene
  Interventions: Procedure: Interrupted subcuticular skin closure

INTERVENTIONS:
Procedure: Interrupted subcuticular skin closure — skin is closed with interrupted mattress subcuticular sutures using non-absorbable polypropylene after elective cesarean section
  Arms: Interrupted subcuticular
Procedure: continuous subcuticular skin closure — skin is closed with continuous subcuticular sutures using non-absorbable polypropylene after elective cesarean section
  Arms: continous subcuticular

SUMMARY:
Non-diabetic pregnant women who undergo elective CS will be randomized into two groups: group I included women who has their skin closed with subcuticular interrupted mattress suture using non-absorbable polypropylene, and group II included women who has their skin closed with subcuticular continous suture using the same suture material

DETAILED DESCRIPTION:
Non-diabetic pregnant women who undergo elective CS will be randomized into two groups: group I included women who had their skin closed with subcuticular interrupted mattress suture using non-absorbable polypropylene, and group II included women who had their skin closed with subcuticular continous suture using the same suture material.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Overall good health
* Elective Cesarean section ASA class 1 or 2

Exclusion Criteria:

* Allergy to synthetic suture materials
* Diabetes whether gestational or pregestational
* use of steroid or immunosuppresive medication within last 6 month of procedure
* Skin sepsis or systemic fever
* BMI > 35
* History of keloid or hypertrophic scar formation or dermatologic conditions known to impair wound healing ASA class 3 or 4

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 169 (Actual)
Dates: Start 2017-04-16 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
wound infection | 10 days after surgery
  occurrence of signs of wound infection

SECONDARY OUTCOMES:
scar dehiscence | 10 days after surgery
  occurrence of scar dehiscence or incisional hernia
wound seroma | 10 days after surgery
  occurrence of seroma of wound
the need for reclosure | 10 days after surgery
  actual gapping of wound
postoperative pain | 12 hours after surgery
  through visual analogue score The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
wound hematoma | 10 days after surgery
  occurrence of subcutanous hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes